CLINICAL TRIAL: NCT00427089
Title: Parallel Group Comparison of the New 2 Liter Gut Cleansing Solution NRL 994 Versus Sodium Phosphate Preparation in Routine Colon Cleansing Prior to Colonoscopies for Colon Tumor Screening.
Brief Title: Comparison of 2L NRL994 With NaP Preparation in Colon Cleansing Prior to Colonoscopies for Colon Tumor Screening
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Hans-Jürgen Gruss, Norgine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NRL 994-01/2004 (HSG)
Record Dates: First submitted 2007-01-25; First posted 2007-01-26 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Colonoscopy
Keywords: Colon cleansing; Polyethylene Glycol; Sodium Phosphate
MeSH Terms: interventions — MoviPrep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 2L gut cleansing solution
  Interventions: Drug: Macrogol 3350 Na sulphate NaCl KCl Ascorbic Acid Na Ascorbate
- 2 (Active Comparator)
  Interventions: Drug: Sodium Phosphate solution (NaP)

INTERVENTIONS:
Drug: Macrogol 3350 Na sulphate NaCl KCl Ascorbic Acid Na Ascorbate — 2L gut lavage solution
  Other Names: MOVIPREP®
  Arms: 1
Drug: Sodium Phosphate solution (NaP) — 45 ml solution; BID
  Arms: 2

SUMMARY:
To compare the efficacy, acceptability and safety of the new 2 liter gut cleansing solution (Moviprep) and NaP preparation in routine colon cleansing prior to tumor screening colonoscopies

DETAILED DESCRIPTION:
This was a randomized and multicenter phase III study in ambulatory subjects undergoing an elective colonoscopy for colon cancer screening. Gut cleansing was performed using either the 2 liters of Moviprep gut lavage solution or the 90 ml NaP-containing preparation prior to colonoscopy. Efficacy, acceptability and safety assessments was performed.

ELIGIBILITY:
Inclusion Criteria:

1. The subject's written informed consent had to be obtained prior to inclusion.
2. Male or female ambulatory subjects with an age of 18 to 85 years planned to undergo a complete colonoscopy for colon cancer screening
3. Willing, able and competent to complete the entire procedure and to comply with study instructions
4. Females of childbearing potential had to employ an adequate method of contraception

Exclusion Criteria:

1. Ileus
2. Intestinal obstruction or perforation
3. Toxic megacolon
4. History of colonic resection
5. Requirement for permanent medication and associated stable serum concentrations (e.g. neuroleptic drugs)
6. Congestive heart failure (NYHA III + IV)
7. Acute life threatening cardiovascular disease
8. Untreated or uncontrolled arterial hypertension (max. > 170 mmHg and min > 100 mmHg)
9. Known moderate to severe renal insufficiency
10. Severe renal failure
11. Severe liver failure
12. Known glucose 6 phosphatase dehydrogenase deficiency
13. Known phenylketonuria
14. Known hypersensitivity to polyethylene glycols, NaP and/or Vitamin C
15. Concurrent participation in an investigational drug study or participation within 30 days of study entry
16. Females who were pregnant, nursing or planning a pregnancy. Females of child bearing potential not using reliable methods of contraception
17. Subject had a condition or was in a situation, which in the investigators opinion might have put the subject at significant risk, might confound the study results, or might interfere significantly.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2004-09; Study Completion 2005-05

PRIMARY OUTCOMES:
Efficacy was measured as the degree of cleansing using a 5 grades scale for each of the predefined colon areas resulting into a final grading of the overall quality of gut preparation (A or B: "success" versus C or D: "failure").

SECONDARY OUTCOMES:
the "overall" judgment of the investigator for the colon preparation was documented.
Subject satisfaction/acceptance with the gut lavage procedure was recorded on a VAS scale ranging from 0 to 100 mm.
The taste of the solutions was assessed.
Acceptability and tolerance for the subject was compared.
All Adverse Events were recorded to evaluate the safety.
Laboratory tests (such as blood chemistry and hematology) were conducted to support the safety data as well as measurement of body weight, blood pressure and pulse rate, but also tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Ell, Prof Dr med, Principal Investigator — Dr. Horst Schmidt Kliniken GmbH
Locations (12):
- Germany (12):
  - Klinikum Aschaffenburg Am Hasenkopf 1, Aschaffenburg, Bavaria
  - Schiessgrabenstr. 34, Augsburg, Bavaria
  - Spardorfer Str. 39, Erlangen, Bavaria
  - Heiligengrabstr. 22, Hof, Bavaria
  - Rätestr. 20, Kirchheim, Bavaria
  - Sternbergstr. 8, Regensburg, Bavaria
  - Israelitische Krankenhaus Abt. innere Medizin Orchideenstieg 14, Hamburg, Hamburg
  - Dieburger Str. 29, Darmstadt, Hesse
  - Unter den Eichen 26, Oldenburg, Lower Saxony
  - Erzbergstr. 113, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Kath. Krankenhaus St. Johann Nepomuk Abt. für Endoskopie Haarbergstr. 72, Erfurt, Thuringia
  - Uferstr. 3, Minden, Westfalen-Lippe

REFERENCES:
- [Result] Ell C, Fischbach W, Layer P, Boehm G, Bokemeyer B, Frick B, et al. Polyethylene Glycol with electrolytes and ascorbic acid versus sodium phosphate for bowel cleansing before coloscopy for cancer screening: a randomised, controlled trial. Endoscopy 2006; 38 (Suppl II): A18
- [Derived] Ell C, Fischbach W, Layer P, Halphen M. Randomized, controlled trial of 2 L polyethylene glycol plus ascorbate components versus sodium phosphate for bowel cleansing prior to colonoscopy for cancer screening. Curr Med Res Opin. 2014 Dec;30(12):2493-503. doi: 10.1185/03007995.2014.960513. Epub 2014 Sep 23. PMID 25180609